CLINICAL TRIAL: NCT00512850
Title: The Nurses' Health Study (NHS) and Health Professionals Follow-Up Study (HPFS) Folic Acid Prevention Trial
Brief Title: Folic Acid in Preventing Colorectal Polyps in Patients With Previous Colorectal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dana-Farber/Brigham and Women's Cancer Center (Other)
Responsible Party: Principal Investigator, Edward Giovannucci, Edward Giovannucci, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BWH-1999-P-001674/10; CDR0000559650 (Registry Identifier: PDQ (Physician Data Query)); BWH-94-06819 (Other: Brigham and Women's Hospital Legacy #); R01CA067883 (NIH)
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Adenoma of Large Intestine
Keywords: Folic acid; Adenoma of Large Intestine
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Folic acid (Other): Folic acid supplement 1g/day
  Interventions: Dietary Supplement: Folic acid
- Placebo (Other): Placebo pill once per day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Folic acid — Intervention group 1g folic acid per day
  Arms: Folic acid
Other: Placebo — One placebo pill per day
  Arms: Placebo

SUMMARY:
RATIONALE: Chemoprevention is the use of certain substances to keep cancer from forming. The use of folic acid may prevent colorectal cancer.

PURPOSE: This randomized clinical trial is studying how well folic acid works compared with a placebo in preventing colorectal polyps in patients who have had previous colorectal polyps.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if folic acid supplementation lowers the adenoma recurrence rate.

Secondary

* Determine the number of adenomas per patient and the size and histology of the adenoma.
* Assess the interaction between folic acid and alcohol, methionine, and aspirin intake.
* Assess the interaction between folic acid and pretrial and midtrial folate levels.
* Assess other complementary biomarkers such as DNA methylation and blood folate level as risk factors for polyp recurrence.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral folic acid once daily.
* Arm II: Patients receive oral placebo once daily. At least 1 year after beginning treatment, patients are sent a blood collection kit in order to measure plasma vitamin B12 levels, to measure folate to assess compliance.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Participated in the Nurses' Health Study (NHS I) or the Health Professionals Follow-Up Study (HPFS) and have had a previous confirmed diagnosis of adenomatous polyp of the colon or rectum
* Plan on having an endoscopy within 4 years after initiation of the trial
* Must release medical records regarding past and any future endoscopies

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Plasma vitamin B12 concentration of ≥ 300 pg/mL or have a vitamin B12 concentration between 200 and 299 pg/mL and a methylmalonic acid (MMA) level ≤ 32 µg/L

Exclusion criteria:

* Diagnosis of cancer other than non-melanoma skin cancer, or early stage breast or prostate cancer
* Diagnosis of homocystinemia
* Diagnosis of pernicious anemia
* Any gastrointestinal disorder that could lead to a vitamin B12 deficiency
* Diagnosis of cirrhosis or pancreatitis
* Diagnosis of epilepsy, Alzheimer's disease, Parkinsonism, and psychiatric disorders that may interfere with normal functioning

PRIOR CONCURRENT THERAPY:

Exclusion criteria:

* No prior gastrectomy, total colectomy, or pancreatectomy
* Other concurrent multivitamins or supplements that contain folic acid (they may take specific supplements, such as A, C, E, calcium, and iron, or antioxidant formula vitamins)
* No concurrent methotrexate or anticonvulsant

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 1996-05; Primary Completion 2004-03 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Recurrent colorectal adenoma | May 1996-March 2004

SECONDARY OUTCOMES:
recurrent adenoma by location, size, stage, number, | May1996-March 2004

CONTACTS AND LOCATIONS:
Overall Officials: Edward L. Giovannucci, MD, ScD, Principal Investigator — Dana-Farber/Brigham and Women's Cancer Center

REFERENCES:
- [Result] Wu K, Platz EA, Willett WC, Fuchs CS, Selhub J, Rosner BA, Hunter DJ, Giovannucci E. A randomized trial on folic acid supplementation and risk of recurrent colorectal adenoma. Am J Clin Nutr. 2009 Dec;90(6):1623-31. doi: 10.3945/ajcn.2009.28319. Epub 2009 Oct 28. PMID 19864409
- [Result] Figueiredo JC, Mott LA, Giovannucci E, Wu K, Cole B, Grainge MJ, Logan RF, Baron JA. Folic acid and prevention of colorectal adenomas: a combined analysis of randomized clinical trials. Int J Cancer. 2011 Jul 1;129(1):192-203. doi: 10.1002/ijc.25872. Epub 2011 Apr 1. PMID 21170989